CLINICAL TRIAL: NCT06111833
Title: Optimized Diagnosis and Precision Medicine of MODY (Maturity-Onset Diabetes of the Young)
Brief Title: Optimized Diagnosis and Precision Medicine of MODY
Status: Recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: CF23186B
Record Dates: First submitted 2023-10-04; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Maturity-Onset Diabetes of the Young (MODY); Type 2 Diabetes; Diabetes Complications
MeSH Terms: conditions — Mason-Type Diabetes; Diabetes Mellitus, Type 2; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples will also be collected for biochemical tests and genetic tests
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case (MODY): 1. Age at diagnosis of diabetes ≤ 25 years old; and
  2. BMI ≤ 25kg/m2; and
  3. At least one parent suffers from type 2 diabetes
- Family: Direct blood relatives/brothers and sisters of the Case group, who have contacted the research team through the subjects and are willing to participate in this study after giving full informed consent.
- Control: 1. Age at diagnosis of diabetes ≤ 40 years old, and without typical MODY characteristics
  2. At least one parent suffers from type 2 diabetes

SUMMARY:
The goal of this observation is to establish a complete registry for the clinical manifestations, environment, genetic, and other related gene variation information of young-onset diabetic patients. Moreover, according to the physiological and pathological mechanisms of different genes, the impact on the clinical characteristics of diabetes, the therapeutic response to drugs, and the impact on complications will be analyzed.

The main questions are:

1. The distribution of different types of MODY
2. The phenotypes and clinical characteristics of different types of MODY
3. Response to antidiabetic drugs among different types of MODY

Once the participant is enrolled, their questionnaire information (including disease course and development, health history, family history, drug history, etc.), medication, outpatient/inpatient medical history, etc. will be collected and logged in. Blood and urine samples will also be collected for biochemical tests genetic testing, etc.

At the same time, the investigators will conduct a continuous follow-up on a regular basis (3 months, 6 months, 12 months, 24 months, and 5 years after the study subject is enrolled).

Young-onset type 2 diabetes will be compared to see the difference in clinical presentations and responses to antidiabetic drugs.

DETAILED DESCRIPTION:
Diabetes and its complications rank among the top ten death causes in Taiwan. In Taiwan, besides the high prevalence, diabetes also shows a trend in younger people. Compared with type 2 diabetes which typically develops at older ages, young-onset diabetes (YOD) has a faster decline in the function of islet cells and a higher risk of complications. These young-onset diabetic patients may belong to different subtypes, and each subtype has different clinical manifestations or genetic characteristics, while the physiological and pathological mechanisms behind them are very complex and closely affect the subsequent treatment decisions. Among young-onset diabetes, maturity-onset diabetes of the young (MODY) has the most obvious genetic predisposition and family history. If the diagnosis is confirmed, it may be possible to directly target the unique defect of the relevant gene and accurately select the appropriate drug therapy to help patients achieve good blood sugar control as soon as possible. This five-year proposal is aimed to target 1,500 young-onset diabetic patients (case group) as well as 500 young-onset, but not MODY, diabetic patients (control group). Once the study subject is enrolled, their questionnaire information (including disease course and development, health history, family history, drug history, etc.), medication, outpatient/inpatient medical history, etc. will be collected and logged in. Blood and urine samples will also be collected for biochemical tests genetic testing, etc. At the same time, the investigators will conduct a continuous follow-up on a regular basis (3 months, 6 months, 12 months, 24 months, and 5 years after the study subject is enrolled). The aim of this proposal is to establish a complete registry for the clinical manifestations, environment, genetic, and other related gene variation information of young-onset diabetic patients. Moreover, according to the physiological and pathological mechanisms of different genes, the impact on the clinical characteristics of diabetes, the therapeutic response to drugs, and the impact on complications will be analyzed. It is expected that different subtypes of early-onset diabetes can be established for genetic counseling, prevention, health education, and treatment selection strategies to achieve good blood sugar and other metabolic control in time, so as to achieve individualized precision medical prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Case Group Diagnosis of diabetes at or before 25 years of age. BMI (Body Mass Index) of 25 kg/m² or lower. Having at least one parent diagnosed with type 2 diabetes.
2. Family Group Direct blood relatives of the case group, including brothers and sisters of the case group, who have contacted the research team through the subjects.

   Expressing willingness to participate in this study after granting informed consent.
3. Control Group Diagnosis of diabetes occurred at or before the age of 40, and the individual lacks typical MODY (Maturity-Onset Diabetes of the Young) characteristics.

At least one parent has been diagnosed with type 2 diabetes.

Exclusion Criteria:

1. Confirmed Diagnosed with type 1 diabetes.
2. Under 18 years of age.
3. Unable to personally provide informed consent.
4. Patients with unrelieved leukemia.
5. Patients who have undergone chemotherapy or radiation therapy for cancer within the last 12 months.
6. Cases that have received a blood transfusion within the last six months.
7. Unwilling or unable to continue treatment follow-up at this hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with young-onset diabetes who receive regular follow-ups at TCVGH and provide informed consent after fully understanding the study's requirements.
  Additionally, direct blood relatives of the case group, including brothers and sisters, who have contacted the research team through the subjects, and have expressed their willingness to participate in this study after granting informed consent
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2028-04-21 (Estimated); Study Completion 2028-05-21 (Estimated)

PRIMARY OUTCOMES:
Glucose control | 3 months
  serum concentration of Fasting glucose (mg/dl) HbA1C (%)
Genetic testing for evaluate the different types of MODY | 1 year
  Genotype evaluate by WES: Pathogenic or likely pathogenic Vairants rate (%)

SECONDARY OUTCOMES:
Renal function | 3 months
  Concentration of urine albumin-creatinine ratio: UACR (mg/g); Serum creatinine mg/dL
Sudomotor function | 1 year
  value of Electrochemical Skin Conductance: μS

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jing Sheen, MD. PHD, Principal Investigator — Division of Endocrinology and Metabolism in Taichung Veterans General Hospital
Locations (1):
- Taichung veterans general hospital, Taichung, Taiwan